CLINICAL TRIAL: NCT04049448
Title: A Follow-up Phase 2a Open-label Study to Evaluate the Long-term Safety and Efficacy Profile of ABX464 in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Study Evaluating the Long-Term Safety and Efficacy of ABX464 in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-302
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate to severe Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Open-label, follow-up study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABX464 50 mg (Experimental): All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 2 years (104 weeks)
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 2 years (104 weeks).

SUMMARY:
A phase 2a open-label study to evaluate the long-term safety and efficacy of ABX464 50mg as maintenance therapy in patients with moderate to severe rheumatoid arthritis.

DETAILED DESCRIPTION:
This Phase 2a open-label study aims at investigating the long-term safety and efficacy of an oral dose of ABX464 in patients who have been previously enrolled in the ABX464-301 clinical study and who are willing to continue their treatment.

All patients will receive ABX464 given at 50mg o.d. irrespectively of their previous treatment received in the ABX464-301 study (i.e. ABX464 or Placebo).

The enrolment in this follow-up study will be based on the willingness of the subject to carry on his/her participation and also based on investigator's judgement.

Patients will be treated with ABX464 for a period of 52 weeks. If they achieve a clinical response on Week 52 (defined as DAS28-CRP ≤ 2,6 for anti-TNFα naïve patients or DAS-28-CRP ≤ 3,2 for patients previously treated by anti-TNFα), they will be eligible to continue treatment for up to 104 weeks.Patients will be followed up at week , week 2 and then, on a monthly basis the first year (up to W52), and quaterly the second year (up to W104).

ELIGIBILITY:
Inclusion Criteria:

* Patients previously enrolled in the ABX464-301 clinical study who have completed the initial 12 weeks of treatment period;

Criteria that should be met by patients at week 52 to be eligible for 52 additional weeks of study treatment:

▪ Patients should be in clinical response. Clinical response is defined as: DAS28-CRP ≤ 2,6 for anti-TNFα naïve patients or DAS-28-CRP ≤ 3,2 for patients previously treated by anti-TNFα.

Exclusion Criteria:

* Any condition, which in the opinion of the investigator, could compromise the patient's safety or adherence to the study protocol

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in the ABX464 treated Patients, categorized by severity | through study completion (average of 104 weeks)
  Incidence of adverse events emerging during the treatment

SECONDARY OUTCOMES:
Proportion of patients achieving Low Disease Activity (LDA) | Week 4, Week 12, Week 24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  Low Disease Activity (LDA) is defined as DAS28-ESR <=3.2
Proportion of patients achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean remission | Week 4, Week 12, Week24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  The ACR/EULAR boolean-based remission is a validated criteria based on: Tender/painful Joint Count (28), Swollen Joint Count (28), C-Reactive Protein, patient global assessment of disease, All ≤ 1
Proportion of patients achieving Simplified Disease Activity Score (SDAI) remission | Week 4, Week 12, Week 24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  The SDAI remission is considered achieved if the SDAI score ≤ 3.3
Proportion of patients achieving Clinical Disease Activity (CDAI) remission | Week 4, Week 12, Week 24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  The CDAI remission is considered achieved if the CDAI score ≤ 2.8
Proportion of patients achieving ACR20/50/70 response | Week 4, Week 12, Week 24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  The categorical American College of Rheumatology 20% or 50% or 70% (ACR20/50/70) response is a validated index of rheumatoid arthritis disease activity, defined by the number of patients who achieved at least 20% or 50% or 70% improvement in the ACR response.
Proportion of patients achieving categorical Disease Activity Scores (DAS) (measured on 28 joints) - C-Reactive Protein (DAS28-CRP) response | Week 4, Week 12, Week 24, Week36, Week 52, Week 65, Week 78, Week 91 and Week 104
  Proportion of patients achieving categorical Disease Activity Score (DAS) DAS28-C-Reactive Protein (CRP) [DAS28-CRP] response will be measured as moderate/good European League Against Rheumatism (EULAR) response
Time to onset of the Low Disease Activity (LDA) remission | up to 104 weeks
  time when DAS28-ESR <=3.2
Time to onset of the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean remission | up to 104 weeks
  The ACR/EULAR remission is a validated criteria based on: Tender/painful Joint Count (28), Swollen Joint Count (28), C-Reactive Protein, patient global assessment of disease, All ≤ 1.
  Time to onset will be when this criteria will be ≤ 1

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Desroys du Roure, PharmD, Study Chair — Abivax S.A.
Locations (14):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
- France (3):
  - CHU de Brest - Hôpital Cavale Blanche, Brest
  - CHU DE MONTPELLIER - Hôpital Lapeyronie, Montpellier
  - CHR d'Orléans, Orléans
- Hungary (3):
  - Complex Medical Centre - Déli Klinika, Budapest
  - CRU Hungary Ltd., Miskolc
  - CMed Rehabilitációs és Diagnosztikai Központ, Székesfehérvár
- Poland (6):
  - ClinicMed Daniluk, Nowak Sp. J., Bialystok
  - Pratia MCM, Krakow
  - Zespół Poradni Specjalistycznych REUMED, Lublin
  - NZOZ Lecznica MAK-MED S.C., Nadarzyn
  - Medyczne Centrum Hetmańska, Poznan
  - National Institute of Geriatrics, Warsaw

IPD SHARING:
Plan to Share IPD: No